CLINICAL TRIAL: NCT05859451
Title: Evaluation of Tobacco Heating System (THS) Compared to Conventional Cigarette Smoking During the Closed Lower Limb (Tibia and Femur) Fracture Healing in Orthopedic Smokers' Patients
Brief Title: Effect of Tobacco Heating System (THS) on Closed Lower Limb Fracture Healing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Philip Morris Products S.A. (Industry)
Responsible Party: Principal Investigator, Prof. Dr. rer. nat. Andreas Nüssler, Profesor Doctor, University Hospital Tuebingen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIS.SWI-THS.2022
Record Dates: First submitted 2023-03-30; First posted 2023-05-16 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Smoking; Tibia Fracture
Keywords: Bone healing; Tobacco heating system; Smoking cessation
MeSH Terms: conditions — Smoking; Tibial Fractures; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Smokers (No Intervention): Participants subject to an orthopedic surgery (does not want to quit smoking conventional cigarettes) will continue smoking conventional cigarettes ad libitum for a period of 6 month post surgery
- Smokers willing to switch to THS (Experimental): Participants subject to an orthopedic surgery (currently smoking conventional cigarettes) will start to used THS ad libitum for a period of 6 month post surgery
  Interventions: Device: Tobacco Heating System (THS)
- Ex Smokers (Active Comparator): Participants subject to an orthopedic surgery will not smoke cigarettes or use electronic nicotine deliver systems for a period of 6 month post surgery
  Interventions: Other: Smoking abstinence

INTERVENTIONS:
Device: Tobacco Heating System (THS) — Participant who are not willing to quit cigarette smoking during the study duration will switch from cigarettes to using THS
  Other Names: IQOS 3 DUO
  Arms: Smokers willing to switch to THS
Other: Smoking abstinence — Participant who are willing to quit cigarette smoking and will not use any electronic nicotine delivery system during the study duration
  Arms: Ex Smokers

SUMMARY:
The goal of this clinical trial is to investigate the role of switching from cigarette smoking (CS) to tobacco heat system (THS) on the clinical outcome of closed lower limb (tibia and femur) fractures from smokers' orthopedic patients. Validated and standardized assays, medical state and self-reported outcomes will be evaluated in orthopedic patients' smokers or switch from CS to using THS throughout six months compare to ex-smokers (control).

ELIGIBILITY:
Inclusion Criteria:

* Closed tibia or femur fracture (according to AO/OTA: 41A2-41C3, 42A-C, 43A-C, 32A-C, 33A2-3, 33B-C) which is surgically treated within 14 days after the trauma at the BG trauma clinic Tübingen.

Additional inclusion criteria for the smoking and THS groups:

* Smokers with 10-20 packyears smoking history.
* Smoking history >10 years.
* Decision not to participate in the free smoking cessation seminars.

Exclusion Criteria:

* Legal guardian or loss of capacity to consent.
* Refusal to participate in the study.
* Open fractures or concomitant injuries or complications requiring surgery existing at the time of surgical indication.
* Initial surgical treatment of the fracture has occurred ex domo.
* No initial surgical treatment within 14 days of sustained trauma.
* Using nicotine delivery electronic devices.
* Pre-existing autoimmune, immunological, bone or malignant diseases.
* Pregnant, breastfeeding and women of childbearing age with existing desire to have children.
* History of alcohol abuse or drug abuse.
* Taking antioxidants approval by the German Federal Institute for Drugs and Medical Devices (BfArM).
* Taking drugs with known effect on bone metabolism (according to Institute for medical and pharmaceutical examination issues (IMPP): allosteric CaSR modulators, bisphosphonates, calcium release inhibitors, alkaline earth ions, RANKL inhibitors, calcitriol, colecalciferol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-04-17 (Estimated)

PRIMARY OUTCOMES:
Concentration of Procollagen Type 1 N-Terminal Propeptide (CICP) | 6 months after tibia fracture surgery
  Marker collagen formation - bone formation

SECONDARY OUTCOMES:
Concentration of Alkaline Phosphatase (BAP) | 6 months after tibia fracture surgery (time points: approx. one week pre-, six weeks post-, twelve weeks post- and six months post-surgery)
  Marker osteoblast activity
Concentration of Osteoprogesterin | 6 months after tibia fracture surgery (time points: approx. one week pre-, six weeks post-, twelve weeks post- and six months post-surgery)
  Decoy receptor RANKL - inhibit osteoclast differentiation
Concentration of Osteopontin | 6 months after tibia fracture surgery (time points: approx. one week pre-, six weeks post-, twelve weeks post- and six months post-surgery)
  Extracellular structural protein and an organic component of bone - favors osteoclast adherence
Concentration of N-terminal telopeptide (NTx) | 6 months after tibia fracture surgery (time points: approx. one week pre-, six weeks post-, twelve weeks post- and six months post-surgery)
  Marker collagen degradation - bone resorption
Concentration of Interleukin 1 beta (IL-1β) | 6 months after tibia fracture surgery (time points: approx. one week pre-, six weeks post-, twelve weeks post- and six months post-surgery)
Concentration of Interleukin 6 (IL-6) | 6 months after tibia fracture surgery (time points: approx. one week pre-, six weeks post-, twelve weeks post- and six months post-surgery)
Concentration of Interferon gamma (IFN-γ) | 6 months after tibia fracture surgery (time points: approx. one week pre-, six weeks post-, twelve weeks post- and six months post-surgery)
Concentration of Tumor Necrosis Factor Alpha (TNF-α) | 6 months after tibia fracture surgery (time points: approx. one week pre-, six weeks post-, twelve weeks post- and six months post-surgery)
Number of bridged cortices in conventional X-ray | 6 months after tibia fracture surgery
Number of bridged cortices in computed tomography scan | 6 months after tibia fracture surgery
Bone Stiffness by a CT-based finite element method | 6 months after tibia fracture surgery
  Finite element method will be used to simulate the mechanical behavior (linear-elastic range) of the tibia and predict bending stiffness under a 3-point bending test
Functional index in trauma (FIX-IT) - Score | 6 months after tibia fracture surgery
  Assess weight-bearing and pain in patients with lower extremity fractures eight-bearing and pain in patients with lower extremity fractures. The score rank from 0 to 12 points in 2 domains: the ability to bear weight (maximum 6 points) and pain at the fracture site (maximum 6 points). The scores in both domains, which are weighted equally, are summed to obtain the final total score; (maximum 12 points indicates the highest level of function).
Loading of the injured extremity | 6 months after tibia fracture surgery
  The time period with no, sole contact, partial or full load on the injured extremity.
Lower Extremity Functional Scale (LEFS) - Score | 6 months after tibia fracture surgery
  The Lower Extremity Functional Scale (LEFS) is a questionnaire (20 questions) about a person's ability to perform everyday tasks. The LEFS will be used to evaluate the functional impairment of a patient with a disorder of lower extremity. The score rank from 0 to 80 points. The maximum score (80 point) indicates no functional limitations.
Number of complications associated with the healing process | 6 months after tibia fracture surgery
Number of hospital stay and incapacity to work [days] | 6 months after tibia fracture surgery
Physicians Global Assessment to measure quality of life (PROMIS GH10 v 1.2) - Score | 6 months after tibia fracture surgery
  The Global Health Patient-Reported Outcomes Measurement Information System (PROMIS- 10) scale is a ten-item patient reported measure of physical, mental and social health. Two summary scores are calculated from the results of the questions: a global physical health score and a global mental health score. These scores are then normalized to the general population using the "T-score." The score ranges from 0 to 20 points. 0 points represent the most severe physical and/or mental impairment of the patient, while 20 points represent the best possible health status.
Visual Analog Score for pain (VAS) - Score | 6 months after tibia fracture surgery
  Visual Analog Scale for Pain (VAS) provide an estimate of patients' pain intensity. Scale from cero (no pain) to 10 (extreme pain).

OTHER OUTCOMES:
Concentration of Soluble intercellular adhesion molecule-1 (sICAM-1) | 6 months after tibia fracture surgery (time points: approx. one week pre-, six weeks post-, twelve weeks post- and six months post-surgery)
Concentration of High densitiy lipoprotein cholesterol levels (HDL) | 6 months after tibia fracture surgery (time points: approx. one week pre-, six weeks post-, twelve weeks post- and six months post-surgery)
Concentration of Leucocytes | 6 months after tibia fracture surgery (time points: approx. one week pre-, six weeks post-, twelve weeks post- and six months post-surgery)
Concentration of Erythrocytes | 6 months after tibia fracture surgery (time points: approx. one week pre-, six weeks post-, twelve weeks post- and six months post-surgery)
Concentration of Hemoglobin | 6 months after tibia fracture surgery (time points: approx. one week pre-, six weeks post-, twelve weeks post- and six months post-surgery)
Concentration of Thrombocytes | 6 months after tibia fracture surgery (time points: approx. one week pre-, six weeks post-, twelve weeks post- and six months post-surgery)
Mean corpuscular volume | 6 months after tibia fracture surgery (time points: approx. one week pre-, six weeks post-, twelve weeks post- and six months post-surgery)
Hematocrit levels | 6 months after tibia fracture surgery (time points: approx. one week pre-, six weeks post-, twelve weeks post- and six months post-surgery)
Mean corpuscular hemoglobin levels | 6 months after tibia fracture surgery (time points: approx. one week pre-, six weeks post-, twelve weeks post- and six months post-surgery)
Corpuscular hemoglobin concentration | 6 months after tibia fracture surgery (time points: approx. one week pre-, six weeks post-, twelve weeks post- and six months post-surgery)
Protein c reactive levels | 6 months after tibia fracture surgery (time points: approx. one week pre-, six weeks post-, twelve weeks post- and six months post-surgery)
Alcohol consume | 6 months after tibia surgery
  Compensation cigarette abstinence with alcohol
Questionnaire on Smoking Urges (QSU-G) - Score | 6 months after tibia surgery
Smoking behaviour | 6 months after tibia surgery
  Number of cigarettes or THS heets consume
Nicotine withdrawal syndrome assessment - Checklist | 6 months after tibia surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Siegfried Weller Institutes, BG-Trauma Clinic, Department of Traumatology, Eberhard Karls University Tübingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
All IPD (in an anonymous form) that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: 6 months after results are published in peer-reviewed international journal

REFERENCES:
- [Background] Aspera-Werz RH, Ehnert S, Muller M, Zhu S, Chen T, Weng W, Jacoby J, Nussler AK. Assessment of tobacco heating system 2.4 on osteogenic differentiation of mesenchymal stem cells and primary human osteoblasts compared to conventional cigarettes. World J Stem Cells. 2020 Aug 26;12(8):841-856. doi: 10.4252/wjsc.v12.i8.841. PMID 32952862
- [Background] Weng W, Bovard D, Zanetti F, Ehnert S, Braun B, Uynuk-Ool T, Histing T, Hoeng J, Nussler AK, Aspera-Werz RH. Tobacco heating system has less impact on bone metabolism than cigarette smoke. Food Chem Toxicol. 2023 Mar;173:113637. doi: 10.1016/j.fct.2023.113637. Epub 2023 Jan 25. PMID 36708864
- [Background] Moritz Herbst, Romina Aspera-Werz, Benedikt Braun, Kevin Schulz, et al. (2024). Evaluation of the Tobacco Heating System (THS) During Closed Lower Limb Fracture Healing in Trauma Smokers' Patients. Qeios. doi:10.32388/DE0EAE.2.